CLINICAL TRIAL: NCT04150146
Title: A Randomized, Open Label, Single Dose, Crossover Study to Evaluate the Food Effect on the Pharmacokinetics of "Rebamipide Sustained Release (SR) 150mg" in Healthy Volunteers
Brief Title: To Evaluate Food Effect on the Pharmacokinetics of Rebamipide in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 037-402-00036
Record Dates: First submitted 2019-09-30; First posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (RT) (Other): [Sequence A (RT) & Sequence B (TR)] to receive the Investigational Product (IP) by the sequence in each period:
  • Rebamipide SR 150 mg: At 9 am on 1d (8d), take with 150 mL of water under the fasting condition for ≥10 hours or after a high-fat meal.
  Interventions: Drug: Rebamipide SR 150mg after high-fat meal; Drug: Rebamipide SR 150mg under fasting condition
- Sequence B (TR) (Other): [Sequence A (RT) & Sequence B (TR)] to receive the Investigational Product (IP) by the sequence in each period:
  • Rebamipide SR 150 mg: At 9 am on 1d (8d), take with 150 mL of water under the fasting condition for ≥10 hours or after a high-fat meal.
  Interventions: Drug: Rebamipide SR 150mg after high-fat meal; Drug: Rebamipide SR 150mg under fasting condition

INTERVENTIONS:
Drug: Rebamipide SR 150mg after high-fat meal — Test Drug
Drug: Rebamipide SR 150mg under fasting condition — Reference Drug

SUMMARY:
This is a randomized, open label, single dose, crossover study to evaluate the food effect on the pharmacokinetics after single oral dose of "rebamipide SR 150 mg" in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who give consent to voluntary participation by signing the informed consent form
2. Healthy adult males aged ≥19 and ≤45 years at screening
3. Subjects with weight ≥50 kg AND body mass index (BMI) ≥18.0 and ≤27.0

Exclusion Criteria:

1. Subjects with hypersensitivity to the active ingredient of the IP or other anti-ulcer agents or history of clinically significant hypersensitivity
2. Subjects with any past history of gastrointestinal diseases which can affect the absorption of the IP
3. Subjects who have participated in other clinical trial and received any other investigational products within 6 months before the expected date of IP administration
4. Subjects who have taken any inducers or inhibitors of drug metabolism enzyme
5. Subjects who have been on diets that may affect the absorption, distribution, metabolism, and excretion of a drug
6. Subjects who donated whole blood within 2 months or underwent apheresis within 1 month prior to obtaining informed consent or who did not agree to prohibit blood donation
7. Smokers who have smoked >10 cigarettes per day within the last 6 months
8. Subjects with any positive result on HBsAg, hepatitis C virus (HCV) Ab, HIV Ab, and (venereal disease research laboratory) VDRL tests

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2019-07-14 (Actual); Study Completion 2019-07-24 (Actual)

PRIMARY OUTCOMES:
Cmax | From Period1/ Day1 to Period2/Day9
  Peak Plasma Concentration of Rebamipide
AUClast of Rebamipide | From Period1/ Day1 to Period2/Day9
  Area Under the plasma concentration versus time curve last of Rebamipide

SECONDARY OUTCOMES:
t1/2 β of Rebamipide | From Period1/ Day1 to Period2/Day9
  Time taken for half the initial dose of Rebamipide administered to be eliminated from the body
Tmax of Rebamipide | From Period1/ Day1 to Period2/Day9
  Time at which the Cmax of Rebamipide is observed
AUCinf of Rebamipide | From Period1/ Day1 to Period2/Day9
  Area Under the plasma concentration versus time curve inifinite of Rebamipide

CONTACTS AND LOCATIONS:
Locations (1):
- CHA Bundang Medical Center, CHA University, Bundang, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No